CLINICAL TRIAL: NCT05122299
Title: The Effect of coenzymeq10/Collagen Hydrogel on Bone Regeneration in Extraction Socket Prior to Implant Placement in Type ii Diabetic Patients (A Randomized Controlled Clinical Trial)
Brief Title: the Effect of coenzymeq10/Collagen Hydrogel on Bone Regeneration in Extraction Socket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: implants_20_21
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Negative control group (Other)
  Interventions: Procedure: Negative control group
- Positive control group (Active Comparator)
  Interventions: Procedure: Postive control
- Study group (Experimental)
  Interventions: Procedure: Study group

INTERVENTIONS:
Procedure: Negative control group — No intervention after extraction then delayed implant insertion at the site of extraction after three months
  Arms: Negative control group
Procedure: Postive control — Application of collagen only in the socket after extraction then delayed implant insertion at the site of extraction after three months.
  Arms: Positive control group
Procedure: Study group — Application of acombination of CoQ10 and collagen hydrogel in the socket after extraction then delayed implant insertion at the site of extraction after three months.
  Arms: Study group

SUMMARY:
To investigate the effect of CoQ10 in soft tissue healing and bone regeneration after extraction in diabetic patients seeking dental implants. Methods: This study will be a randomized controlled clinical trial, 18 patients will be divided equally into three groups. In-vitro studies will be performed to investigate the release of CoQ10 from collagen, swelling ratio, and evaluation of gelation behavior. The patients will undergo tooth extraction and filling of the socket with either collagen or CoQ10/collagen. Empty sockets will serve as a negative control. The bone regeneration of the socket will be determined by radiography, histology, histomorphometry, and polymerase chain reaction (PCR) for bone markers.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60 years including both males and females .
* Controlled Type II diabetic patients glycosylated hemoglobin (HbA1C) levels less than 7
* Good oral hygiene
* No history of bruxism/ para-functional habits
* Patients accept to sign the informed consent .
* Single or multiple Mandibular teeth requiring extraction.

Exclusion Criteria:

* Uncontrolled diseases that may contraindicate the surgery.
* Somkers patients.
* Osteoporosis.
* Hypersensitivity.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Soft tissue healing | at 1 week
  Landry index will be used to evaluate the parameters of tissue colour, bleeding response to palpation, presence of granulation tissue, characteristics of the incision margins, and the presence of suppuration. This index assesses wound healing using scores from 1 to 5: a wound with very poor healing receives a score of 1, whereas excellent healing receives a score of 5.
change in bone formation | at baseline, 3 months and 6 months
  Conebeam computed tomography (CBCT) will be taken at 3 different timepoints; immediatly after extraction to measure height and width of alveolar bone, before implant placement to place implant in accurate position and to compare it with first one to measure the changes in bone height and width and finally at loading to evaluate marginal bone loss.
Change in implant stability | at baseline and 3 months
  Osstell instrument (Integration Diagnostics, Goteborg, Sweden) with Smartpeg™ (Integration Diagnostics, Goteborg, Sweden), a transducer suitable for implants will be used to assess stability of implants by RFA. ISQ (implant stability quotient) will be obtained from the measurement results. During measurement, the Smartpeg™ will be placed over the location of implant prosthesis and the Osstell probe will be approximated to it from the buccal, palatal, mesial and distal aspects of the implant giving four ISQ values. A mean ISQ for each implant is then calculated by averaging the four values.
  implant stability quotient or ISQ score in a range of 0-100.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt